CLINICAL TRIAL: NCT03327350
Title: The WASPS Trails:WATCHMAN for Second Prevention of Stroke
Brief Title: WATCHMAN for Second Prevention of Stroke (WASPS)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZJU CT009
Record Dates: First submitted 2017-01-07; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-01

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- WATCHMAN transplantation: This group will receive WATCHMAN device implantation.Device implantation included concomitant antithrombotic medication to facilitate device endothelialization: warfarin and aspirin for 45 days. To assess for device stability, peridevice leaks, and device-related thrombus, transesophageal echo (TEE) imaging was performed at 45 days, 6 months, and 12 months. When the 45-day TEE revealed minimal residual peridevice flow (jet width ≤5 mm) and no device-related thrombus, warfarin will be stopped and replaced by clopidogrel, 75 mg daily, until the 6-month visit, after which only aspirin was continued. If an adequate seal is not obtained or a thrombus is detected, patients continue taking warfarin until an adequate seal is attained or thrombus is resolved before transitioning to aspirin.
  Interventions: Device: WATCHMAN transplantation
- Oral anticoagulant therapy: This group will take oral anticoagulant drugs(warfarin or the new oral anticoagulant drugs like Dabigatran ).
  For patients taking warfarin, international normalized ratio (INR) monitoring wil be performed at least every 2 weeks for 6 months and at least monthly thereafter, targeting an INR between 2 and 3. Follow-up visits occurred twice annually after the first year, with neurological assessments at 12 months and yearly thereafter or whenever a neurological event is suspected.
  Interventions: Drug: Oral anticoagulant drugs

INTERVENTIONS:
Device: WATCHMAN transplantation — WATCHMAN Left Atrial Appendage System is a novel device designed to prevent the embolization of thrombi that may form in the LAA. It is hypothesized that it may prevent ischemic stroke and systemic
  Groups: WATCHMAN transplantation
Drug: Oral anticoagulant drugs — This group will take oral anticoagulant drugs(warfarin or the new oral anticoagulant drugs like Dabigatran ).For patients taking warfarin,international normalizedratio (INR) monitoring wil be performed at least every 2 weeks for 6 months and at least monthly thereafter, targeting an INR between 2 and 3. Followup visits occurred twice annually after the first year,with neurological assessments at 12 months and yearly thereafter or whenever a neurological event is suspected.
  Groups: Oral anticoagulant therapy

SUMMARY:
To evaluate the effects of mechanical left atrial appendage (LAA) closure for secondary prevention of stroke in the patients with nonvalvular atrial fibrillation

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia, affecting an estimated 5 million Chinese. Atrial fibrillation is the primary cardiac abnormality associated with embolic stroke; among patients with AF, there is an annual stroke rate, about 5 times for the same age population in sinus rhythm.

Although warfarin therapy is effective at reducing the risk of stroke, chronic anticoagulation presents problems of safety and acceptability for many patients. Drug and dietary interactions, frequent blood tests, and compliance issues all contribute to difficulties with chronic warfarin therapy. New oral anticoagulant compounds with better therapeutic range and without need for similar monitoring, such as Dabigatran, Rivaroxaban, Apixaban and Edoxaban,have been studied, but there is no direct comparison with left atrial appendage closure(LAAC).

However,the left atrial appendage (LAA) is the major location of thrombi in patients with AF. In patients with nonrheumatic AF and thrombus in the left atrium, the clot was located in the LAA in 90%. And the WATCHMAN Left Atrial Appendage System is a novel device designed to prevent the embolization of thrombi that may form in the LAA. It is hypothesized that it may prevent ischemic stroke and systemic thromboembolism in patients with AF.The PROTECT-Af and PREVAIL trails confirmed this device's efficacy and safety, compared with warfarin, for preventing the combined outcome of stroke,systemic embolism, and cardiovascular death. And the device has been approved by China's FDA.

Stroke is the primary cause of death in China, and recurrence of stroke remains a major public health issue.

This cohort study is designed to evaluate the effects of mechanical left atrial appendage (LAA) closure for secondary prevention of ischemic stroke in the patients with nonvalvular atrial fibrillation in China, compared with medicine approach (Warfarin or NOAC),.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* A history of stroke/transient ischemic attack(TIA) over 3 months;
* Paroxysmal, persistent, or permanent nonvalvular AF;
* 4.2 or more CHA2DS2-VASc risk factors
* Eligibility for long-term anticoagulation with warfarin or new oral anticoagulants.

Exclusion Criteria:

* patent foramen ovale with atrial septal aneurysm
* an atrial septal defect
* mechanical valve prosthesis
* left ventricular ejection fraction less than 30%
* mobile aortic atheromata
* symptomatic carotid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 hospitalized patients over 18 years old with nonvalvular atrial fibrillation will be enrolled consecutively
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-11-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
All stroke (including ischemic and hemorrhagic) and systemic embolism, cardiovascular death (limited to any cardiovascular and unexplained) | 3 years

SECONDARY OUTCOMES:
All the serious complications,including the surgery complications and major bleeding events. | 3 years
All-cause death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD,PhD, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided